CLINICAL TRIAL: NCT06171269
Title: A Prospective Study of Lower Dose Radiation (LO-RADS) for Prostate Cancer Using MRI Dose Mapping to Preserve Quality of Life
Brief Title: Using MRI to Identify Areas to Receive Lower Doses of Radiation Treatment in Men With Prostate Cancerdose Mapping to Preserve Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-1023
Record Dates: First submitted 2023-11-14; First posted 2023-12-14 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation therapy (Experimental): Participants will receive MRI scan before starting Radiation treatment. The results of this scan will be used to identify areas of the prostate to receive low doses of radiation (areas that show no cancer cells seen by the MRI scan).
  Interventions: Radiation: Radiation; Radiation: MRI; Other: Androgen Deprivation Therapy

INTERVENTIONS:
Radiation: Radiation — Radiation to the prostate gland will be given daily (Mon-Friday) for 4 weeks.
Radiation: MRI — The study doctor will use an MRI scan to take pictures of the prostate gland. These images of the prostate gland will let the study doctor know which areas of the prostate contain cancer cells that need to be targeted with higher doses of radiation and which uninvolved areas to target with lower doses of radiation.
Other: Androgen Deprivation Therapy — Treatment of treating physician choice will be given for 6-24 months.

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of using an imaging technique called magnetic resonance imaging (MRI) to decrease radiation dose to the uninvolved prostate (areas of the prostate that do not clearly have cancer cells) while increasing radiation dose to the nodules (hardened areas of the prostate that have cancer cells).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) male patients with an ECOG Performance Status 0-2
* Histologically-confirmed, MRI-visible prostate adenocarcinoma with NCCN intermediate- or high-risk disease1 without extra-pelvic metastasis.

Exclusion Criteria:

* Distant metastases
* Prior active treatment for prostate cancer including radical prostatectomy, high-intensity focused ultrasound (HIFU), cryosurgery, ADT, or cytotoxic chemotherapy for treatment of prostate cancer. Patients with prostate cancer on active surveillance prior to the study are not excluded if they have not received active treatment.
* Prior pelvic radiotherapy including brachytherapy.
* Additional active concurrent malignancies (except localized cutaneous squamous or basal cell carcinomas).
* Comorbid conditions that, in the opinion of the treating radiation oncologist, preclude the patient from safely receiving the protocol-specified treatment including RT and/or ADT.
* Patients with contraindications to MRI including patients with ferromagnetic materials in their body (e.g. bioimplants, surgical hardware, shrapnel), patients who are unable to receive contrast due to history of allergy or impaired renal function (glomerular filtration rate < 30 mil/min), and patients unable to tolerate MRI for other reasons (e.g. significant claustrophobia).
* Patients for whom hydrogel or hyaluronic acid spacer will be placed.
* Patients incapable of giving informed consent.
* Patients who are unable to adhere to the experimental protocols for any reason.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be limited to male patients given that prostate cancer does not occur in females.
Enrollment: 60 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2027-02-14 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Improvement in bowel related quality of life | 12 months after treatment
  Decrease by at least 5 points in bowel related endpoints as measured by Expanded Prostate Cancer Index Composite 26 (EPIC-26) questionnaire.

SECONDARY OUTCOMES:
Biochemical control | 2 year after start of treatment
  Number of participants that have failed ADT therapy after 2 years as shown by prostate specific antigen (PSA) levels..
Relationship between Imaging findings and Pathologic (tissue) findings | 12 months post treatment
  Correlation between signs of cancer as seen by imaging and tissue (pathology)
Treatment Side effects | 12 months post treatment
  Number of gastrointestinal, genitourinary, and sexual side effects that are grade 2 or above per the Common Terminology Criteria for Adverse Events (CTCAE)
Patient reported quality of life | 12 months post treatment
  Improvement in patient reported quality of life (shown higher scores of worse symptoms) with the scale values assigned to each question ranging from 0 (best) to 4 (worst) of gastrointestinal, genitourinary, and sexual function as assess by Expanded Prostate Cancer Index (EPIC) questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Liauw, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No